CLINICAL TRIAL: NCT01283477
Title: Efficacy of Acupuncture for Prophylaxis of Intrathecal Morphine Induced Pruritis in Patients Undergoing Caesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Letterkenny General Hospital (Other Government)
Responsible Party: DR. KARTHIK GANESH RAMAMOORTHY , PRINCIPAL INVESTIGATOR, Letterkenny General Hospital, HSE IRELAND
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ITM - LI 11
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2011-01

CONDITIONS: Acupuncture; Morphine Induced Pruritis
Keywords: Caesarean Delivery; Pruritis; Intrathecal Morphine; Acupuncture At LI11
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACUPUNCTURE (Experimental)
  Interventions: Device: ACUPUNCTURE AT LI11
- SHAM ACUPUNCTURE (Sham Comparator)
  Interventions: Device: SHAM ACUPUNCTURE

INTERVENTIONS:
Device: ACUPUNCTURE AT LI11 — ACUPUNCTURE AT LI11 FOR 30 MINUTES PRIOR TO INTRATHECAL MORPHINE & LEFT IN PLACE FOR 30 MINUTES
  Arms: ACUPUNCTURE
Device: SHAM ACUPUNCTURE — SHAM ACUPUNCTURE AT A POINT 2 CM LATERAL TO LI11 30 MINUTES PRIOR TO INTRATHECAL MORPHINE & LEFT IN PLACE FOR 30 MINUTES
  Arms: SHAM ACUPUNCTURE

SUMMARY:
Intrathecal morphine is commonly used for pain relief in caesarean delivery. Side effects such as itch (pruritis) and nausea & vomiting are common and have been shown to be the most common cause for dissatisfaction. The incidence of pruritis is 74% even with current available medications. Acupuncture has been shown to be effective for morphine related side effects but has not been evaluated for prophylaxis of itch in pregnant population.

PRIMARY OBJECTIVE:

Acupuncture at LI 11 reduces the incidence of pruritis after elective caesarean section under spinal with intrathecal morphine

ELIGIBILITY:
Inclusion criteria:

* ASA I & II patients undergoing elective caesarean delivery under spinal with intrathecal morphine

Exclusion criteria:

* Patient refusal
* ASA III & IV patients
* Pre-existing pruritis
* Eczema
* Bleeding tendencies
* Known allergy to any of medications used
* Any contra indication to spinal anaesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pruritis | First 24 hr post intrathecal morphine
  To determine acupuncture at li 11 reduces the incidence of pruritis after elective caesarean delivery under spinal anaesthesia with intrathecal morphine

SECONDARY OUTCOMES:
Severity of pruritis | 1, 4, 8, 24 hr post intrathecal morphine
  To determine acupuncture reduces:
  1. Severity of pruritis
  2. Requirement of relief medications

CONTACTS AND LOCATIONS:
Overall Officials: KARTHIK G RAMAMOORTHY, MBBS, DA,DAc,FCARCSI, Principal Investigator — Letterkenny General Hospital
Locations (1):
- Letterkenny General Hospital, Letterkenny, Donegal, Ireland

REFERENCES:
- [Background] Jiang YH, Jiang W, Jiang LM, Lin GX, Yang H, Tan Y, Xiong WW. Clinical efficacy of acupuncture on the morphine-related side effects in patients undergoing spinal-epidural anesthesia and analgesia. Chin J Integr Med. 2010 Feb;16(1):71-4. doi: 10.1007/s11655-010-0070-7. Epub 2010 Feb 4. PMID 20131040
- [Background] Che-Yi C, Wen CY, Min-Tsung K, Chiu-Ching H. Acupuncture in haemodialysis patients at the Quchi (LI11) acupoint for refractory uraemic pruritus. Nephrol Dial Transplant. 2005 Sep;20(9):1912-5. doi: 10.1093/ndt/gfh955. Epub 2005 Jun 28. PMID 15985509
- [Background] Bonnet MP, Marret E, Josserand J, Mercier FJ. Effect of prophylactic 5-HT3 receptor antagonists on pruritus induced by neuraxial opioids: a quantitative systematic review. Br J Anaesth. 2008 Sep;101(3):311-9. doi: 10.1093/bja/aen202. Epub 2008 Jul 7. PMID 18611915